CLINICAL TRIAL: NCT04925180
Title: Study to Evaluate Physician Awareness and Knowledge of Safety and Safe Use Information for Androcur and Other Cyproterone Acetate Monotherapies in Europe: an Observational Post-Authorisation Joint Safety Study (Safe-CAM)
Brief Title: A Study to Learn About the Awareness and Knowledge That Doctors Have About the Safety and Safe Use Information for Androcur and Other Cyproterone Acetate Treatments in Europe
Acronym: Safe-CAM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21490
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Signs of Androgenisation in Women, e.g. Hirsutism, Androgenetic Alopecia, Acne and Seborrhea; Hypersexuality in Men; Sexual Deviations in Men; Prostate Cancer
Keywords: Cyproterone acetate monotherapies; Effectiveness of risk minimization measures; Survey
MeSH Terms: conditions — Alopecia; Acne Vulgaris; Dermatitis, Seborrheic; Prostatic Neoplasms | interventions — Cyproterone Acetate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: Physicians who have recently prescribed (e.g., within previous 12 months) CPA monotherapy will be invited to complete a brief web-based questionnaire regarding their knowledge of the revised summary of product characteristics (SmPC) and the direct healthcare professional communication (DHPC).
  Interventions: Drug: Cyproterone Acetate (Androcur, BAY94-8367)

INTERVENTIONS:
Drug: Cyproterone Acetate (Androcur, BAY94-8367) — As prescribed by the treating physician

SUMMARY:
Androcur is a type of treatment called cyproterone acetate (CPA). Androcur and other CPA treatments work by blocking a group of male sex hormones called androgens in the body. It can be given to men and women to treat conditions that are caused by higher levels of androgens.

CPAs, including androcur, are currently available as treatments for doctors to give to patients who have these types of conditions. But, in a study, researchers found that participants had a certain medical problem when they took CPAs for a long time. This medical problem was a tumor of the brain or spinal cord that is mostly not malignant and is called meningioma. This eventually led health authorities to change the instructions for how doctors should use CPAs to treat patients. This included what health conditions should be treated with CPAs, how long patients should receive them, and what dose of CPA should be given.

In this study, the researchers want to learn more about how doctors are using CPAs to treat patients after the update to the instructions.

To answer this research question, they will give to the doctors a web-based questionnaire asking about the advisability or necessity of the treatment (also called "indications of approved use"), the measures to be followed to reduce the risk and how much the doctors knew about the risk of meningioma.

The researches will then analyze the answers to the questionnaire. The results will be the percentage of physicians with correct answers for each individual knowledge question from the questionnaire.

The study will include information collected from a diverse sample of doctors during approximately 3 months.

The doctors must have given CPAs as a treatment to at least 1 patient in the last 12 months.

There are no required visits or tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* Licensed and practising dermatologist, endocrinologist, gynaecologist, general practitioners, urologist, oncologist (who treats prostate cancer), or psychiatrist involved in the treatment of hypersexuality/reduction of drive in sexual deviations
* Prescribed CPA monotherapy to at least one patient in the past 12 months
* Work in an office or hospital-based setting
* Electronic acknowledgement of informed consent

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians eligible to participate will include dermatologists, endocrinologists, gynaecologists, general practitioners, urologists, oncologists (who treat prostate cancer), and psychiatrists involved in the treatment of hypersexuality/reduction of drive in sexual deviations who have prescribed CPA in the past 12 months and work in an office or hospital-based setting.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of physicians responding correctly to the knowledge question: The occurrence of meningiomas (single and multiple) in association with CPA monotherapy doses ≥ 25 mg/day | Baseline
Percentage of physicians responding correctly to the knowledge question: Restriction of use of CPA monotherapy 10 mg/50 mg in women when no results have been achieved at lower dose CPA-containing products or with other treatment options | Baseline
Percentage of physicians responding correctly to the knowledge question: Restriction of use of high-dose CPA in men with sexual deviations when other interventions are not appropriate | Baseline
Percentage of physicians responding correctly to the knowledge question: After clinical improvement with CPA monotherapy is achieved, treatment should be maintained with the lowest possible dose | Baseline
Percentage of physicians responding correctly to the knowledge question: The risk of meningioma increases with increasing cumulative doses of CPA | Baseline
Percentage of physicians responding correctly to the knowledge question: CPA is contraindicated in patients with a meningioma or a history of meningioma | Baseline
Percentage of physicians responding correctly to the knowledge question: If a patient treated with CPA monotherapy is diagnosed with meningioma, treatment with all cyproterone-containing products must be permanently stopped | Baseline
Percentage of physicians responding correctly to the knowledge question: Awareness of signs and symptoms of meningiomas | Baseline

CONTACTS AND LOCATIONS:
Locations (5):
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Netherlands
- Many Locations, Multiple Locations, Poland
- Many Locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.